CLINICAL TRIAL: NCT05385783
Title: A Phase I/IIa, Randomized, Double-Blind, Placebo-Controlled Study With an Open-Label Relative Bioavailability and Food Effect Cohort to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of CYB003 in Healthy Participants With and Without Major Depressive Disorder (MDD)
Brief Title: A Study of a Psilocybin Analog (CYB003) in Healthy Participants With and Without Major Depressive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cybin IRL Limited (Industry)
Collaborators: Clinilabs Drug Development Corporation (Unknown); Drug Safety Navigator (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYB003-001
Record Dates: First submitted 2022-05-10; First posted 2022-05-23 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Psilocybin; Psychedelic; Psilocin; CYB003; CYB003-001; Depression; Healthy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A: MDD Participants - CYB003 in 2 of 2 Medicine Sessions (Experimental): Arm A MDD participants will receive CYB003 in 2 of 2 medicine sessions, approximately three weeks apart. The CYB003 dose received will depend on the cohort/time of enrollment. All MDD participants will receive supportive EMBARK psychotherapy throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychotherapy
- B: MDD Participants - Placebo in Medicine Session 1, CYB003 in Medicine Session 2 (Placebo Comparator): Arm B MDD participants will receive placebo in Medicine Session 1, and approximately three weeks later will receive CYB003 in Medicine Session 2. The CYB003 dose received will depend on the cohort/time of enrollment. All MDD participants will receive supportive EMBARK psychotherapy throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychotherapy; Drug: Placebo
- C: Healthy Volunteers - CYB003 in 2 of 2 Medicine Sessions (Experimental): Arm C healthy volunteers will receive CYB003 in 2 of 2 medicine sessions, approximately one to two weeks apart. The CYB003 dose received will depend on the cohort/time of enrollment. All healthy volunteers will receive psychological support throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychological Support
- D: Healthy Volunteers - Placebo in Medicine Session 1, CYB003 in Medicine Session 2 (Placebo Comparator): Arm D healthy volunteers will receive placebo in Medicine Session 1, and approximately one to two weeks later will receive CYB003 in Medicine Session 2. The CYB003 dose received will depend on the cohort/time of enrollment. All healthy volunteers will receive psychological support throughout the study.
  Interventions: Drug: CYB003; Drug: Placebo; Behavioral: Psychological Support
- E: Healthy Volunteers - CYB003 in 3 of 3 Medicine Sessions (Experimental): Arm E healthy volunteers will receive CYB003 in 3 of 3 medicine sessions, approximately one week apart from each other, to assess bioavailability and food effect. The CYB003 dose received will depend on the safety review committee selection/time of enrollment. All healthy volunteers will receive psychological support throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychological Support

INTERVENTIONS:
Drug: CYB003 — CYB003 is a synthetic psilocybin analog.
Behavioral: Psychotherapy — Manualized psychotherapy (called EMBARK) performed by facilitators
  Arms: A: MDD Participants - CYB003 in 2 of 2 Medicine Sessions; B: MDD Participants - Placebo in Medicine Session 1, CYB003 in Medicine Session 2
Drug: Placebo — Placebo
  Arms: B: MDD Participants - Placebo in Medicine Session 1, CYB003 in Medicine Session 2; D: Healthy Volunteers - Placebo in Medicine Session 1, CYB003 in Medicine Session 2
Behavioral: Psychological Support — Manualized psychological support performed by facilitators
  Arms: C: Healthy Volunteers - CYB003 in 2 of 2 Medicine Sessions; D: Healthy Volunteers - Placebo in Medicine Session 1, CYB003 in Medicine Session 2; E: Healthy Volunteers - CYB003 in 3 of 3 Medicine Sessions

SUMMARY:
The purpose of this study is to determine the safety and tolerability of ascending oral doses of CYB003 in healthy participants with and without major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria - MDD & Healthy Volunteer Participants:

* Aged between 21 to 65 years, inclusive, at Screening.
* Has a BMI of 18 to 30 kg/m2, inclusive, at Screening.
* Is ≥60 kg.
* Is negative for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test at Screening and at Day -1.
* Provision of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Additional Inclusion Criteria - MDD Participants Only:

* Has a diagnosis of MDD (as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-V] of moderate to severe degree), established through a full psychiatric work up, who are otherwise healthy.
* Has been on a stable dose of antidepressant medication (no more than 50% change) in the last month prior to Screening and has had an inadequate response, as judged by the Investigator.

Exclusion Criteria - MDD & Healthy Volunteer Participants:

* Clinically significant risk of suicidality, as determined through a comprehensive psychiatric interview.
* Clinically relevant history of abnormal physical health interfering with the study as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including [but not limited to], neurological, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder).
* Diagnosis of hypertension or an arrhythmia.
* History of hypothyroidism and/or current abnormal thyroid function tests.
* Clinically relevant abnormal laboratory results.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Any other concomitant disease or condition that could interfere with, or for which the treatment might interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study.
* Not fluent in the English language.
* Has a presence or relevant history of any of the following medical conditions: organic brain disorders (e.g., epilepsy, seizure, intracranial hypertension, intracranial bleed and aneurysmal disease, brain tumor or other medical conditions associated with seizures or convulsions).
* Positive test for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibody (anti- HCV) or human immunodeficiency virus I and II (anti-HIV I/II) at Screening.
* Has participated in a clinical study and has received a medication or a new chemical entity within 3 months prior to dosing of current study medication.
* Is taking or has taken any drugs known to inhibit monoamine oxidase within 28 days prior to receiving the study drug.
* Is taking or has taken over the counter (OTC) doses of 5-hydroxytrptophan or St John's Wort within 28 days prior to receiving the study drug.
* Donation of blood or plasma of >400 mL within 1 month prior to first dosing until 4 weeks after final dosing.
* Is pregnant, breastfeeding or planning to conceive.
* Known difficulty with obtaining intravenous access.
* Other eligibility considerations (i.e., participant personal circumstances, behavior, and/or any current problem that might interfere with participation or that is incompatible with establishment of rapport or safe exposure to the study drug), as judged by the Investigator.

Additional Exclusion Criteria - Healthy Volunteers Only:

* Current or previously diagnosed with a mental health disorder as defined by DSM-V criteria.
* Use of any prescription medicine (except for hormonal contraceptives, if applicable), certain herbal supplements (to be reviewed by the Investigator), or OTC medicine during the 28 days before dosing.

Additional Exclusion Criteria - MDD Participants Only:

* Current or previous diagnosis of treatment-resistant MDD, defined as failure to respond to 2 or more antidepressant treatments given at an adequate dose for an adequate duration.
* Current or previously diagnosed schizophrenia spectrum or other psychotic disorders, including schizophrenia, schizoaffective disorder, schizotypal disorder, schizophreniform disorder or brief psychotic disorder; current or previous history of bipolar disorder, or current personality disorder.
* Currently receiving a monoamine oxidase inhibitor, tricyclic antidepressant, mirtazapine, an antipsychotic or a mood stabilizer.
* Use of a prescription medicine (except participants may take a stable chronic dose of antidepressant medication(s) and/or sedatives/hypnotics, and may take hormonal contraceptives, if applicable), certain herbal supplements (to be reviewed by the Investigator), or OTC medicine during the 28 days before dosing (some exceptions apply).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Adverse Events (All Arms) | Day 1 thru End of Study Visit (which is: Day 56 Arms A & B; Day 28 Arms C & D; Day 35 Arms E)
  Any untoward medical occurrence in a clinical investigation participant administered a drug and does not necessarily have a causal relationship with the treatment
Resting 12 Lead ECG ventricular rate (Arms A & B) | Screening, Day -1, Day 1, Day 2, Day 21, Day 22, & Day 23
  ventricular rate (beats per minute)
Resting 12 Lead ECG ventricular rate (Arms C & D) | Screening, Day -1, Day 1, Day 2, Day 7, Day 8, & Day 9
  ventricular rate (beats per minute)
Resting 12 Lead ECG ventricular rate (Arms E) | Screening, Day -1, Day1, Day 2, Day 7, Day 8, Day 9, Day 14, Day 15, Day 16
  ventricular rate (beats per minute)
Resting 12 Lead ECG PR interval (Arms A & B) | Screening, Day -1, Day 1, Day 2, Day 21, Day 22, Day 23
  PR interval (milliseconds)
Resting 12 Lead ECG PR interval (Arms C & D) | Screening, Day -1, Day 1, Day 2, Day 7, Day 8, & Day 9
  PR interval (milliseconds)
Resting 12 Lead ECG PR interval (Arms E) | Screening, Day -1, Day1, Day 2, Day 7, Day 8, Day 9, Day 14, Day 15, Day 16
  PR interval (milliseconds)
Resting 12 Lead ECG QRS duration (Arms A & B) | Screening, Day -1, Day 1, Day 2, Day 21, Day 22, Day 23
  QRS duration (milliseconds)
Resting 12 Lead ECG QRS duration (Arms C & D) | Screening, Day -1, Day 1, Day 2, Day 7, Day 8, & Day 9
  QRS duration (milliseconds)
Resting 12 Lead ECG QRS duration (Arms E) | Screening, Day -1, Day1, Day 2, Day 7, Day 8, Day 9, Day 14, Day 15, Day 16
  QRS duration (milliseconds)
Resting 12 Lead ECG QT interval (Arms A & B) | Screening, Day -1, Day 1, Day 2, Day 21, Day 22, Day 23
  QT interval (milliseconds)
Resting 12 Lead ECG QT interval (Arms C & D) | Screening, Day -1, Day 1, Day 2, Day 7, Day 8, & Day 9
  QT interval (milliseconds)
Resting 12 Lead ECG QT interval (Arms E) | Screening, Day -1, Day1, Day 2, Day 7, Day 8, Day 9, Day 14, Day 15, Day 16
  QT interval (milliseconds)
Resting 12 Lead ECG QTcF (Arms A & B) | Screening, Day -1, Day 1, Day 2, Day 21, Day 22, Day 23
  Corrected QT interval by Fredericia (milliseconds)
Resting 12 Lead ECG QTcF (Arms C & D) | Screening, Day -1, Day 1, Day 2, Day 7, Day 8, & Day 9
  Corrected QT interval by Fredericia (milliseconds)
Resting 12 Lead ECG QTcF (Arms E) | Screening, Day -1, Day1, Day 2, Day 7, Day 8, Day 9, Day 14, Day 15, Day 16
  Corrected QT interval by Fredericia (milliseconds)
Holter monitoring (Arms A & B) | Day -1, Day 1, Day 22
  Record of the electrical activity of the heart (Hz)
Holter monitoring (Arms C & D) | Day -1, Day 1, Day 8
  Record of the electrical activity of the heart (Hz)
Holter monitoring (Arm E) | Day -1, Day 1, Day 8, Day 15
  Record of the electrical activity of the heart (Hz)
Columbia Suicide Severity Rating Scale (CSSRS) Lifetime version (All Arms) | Screening
  Evaluation tool that evaluates a lifetime history of suicidal ideation and/or behavior. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of actual attempts are rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care).
Columbia Suicide Severity Rating Scale (CSSRS) Since Last Visit (SLV) (Arms A & B) | Day -1, Day 2, Day 10, Day 17, Day 21, Day 23, Day 31, Day 38, Day 42, and Day 56
  Evaluation tool that evaluates risk for suicide since the last study visit. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of actual attempts are rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care).
Columbia Suicide Severity Rating Scale (CSSRS) Since Last Visit (SLV) (Arms C & D) | Day -1, Day 2, Day 7, Day 9, Day 15, Day 21, Day 28
  Evaluation tool that evaluates risk for suicide since the last study visit. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of actual attempts are rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care).
Columbia Suicide Severity Rating Scale (CSSRS) Since Last Visit (SLV) (Arm E) | Day -1, Day 2, Day 7, Day 9, Day 14, Day 16, Day 21, Day 28, Day 35
  Evaluation tool that evaluates risk for suicide since the last study visit. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of actual attempts are rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care).

SECONDARY OUTCOMES:
Mystical Experience Questionnaire (MEQ30) (Arms A & B) | Day 1 & Day 22
  The revised MEQ30 consists of 30 questions looking back on the entirety of a medicine session, participants are asked to answer each question according to one's feelings, thoughts, and experiences at the time of the session. Each item is rated on a Likert scale (0-None/not at all to 5-Extreme, more than any other time in my life). The minimum score is 0 and the maximum score is 150 with higher scores indicating a greater degree of mystical experience. The MEQ total score is computed by taking the average response to all items.
Mystical Experience Questionnaire (MEQ30) (Arms C & D) | Day 1 & Day 8
  The revised MEQ30 consists of 30 questions looking back on the entirety of a medicine session, participants are asked to answer each question according to one's feelings, thoughts, and experiences at the time of the session. each item rated on a Likert scale (0-None/not at all to 5-Extreme, more than any other time in my life). The minimum score is 0 and the maximum score is 150 with higher scores indicating a greater degree of mystical experience. The MEQ total score is computed by taking the average response to all items.
Mystical Experience Questionnaire (MEQ30) (Arms C & D) | Day 1, Day 8, & Day 15
  The revised MEQ30 consists of 30 questions looking back on the entirety of a medicine session, participants are asked to answer each question according to one's feelings, thoughts, and experiences at the time of the session. each item rated on a Likert scale (0-None/not at all to 5-Extreme, more than any other time in my life). The minimum score is 0 and the maximum score is 150 with higher scores indicating a greater degree of mystical experience. The MEQ total score is computed by taking the average response to all items.
5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC) (Arms A & B) | Day 1 & Day 22
  The 5D-ASC consists of a set of 94 items that participants are asked to rate to what extent the statements apply to one's particular experience, compared to normal waking consciousness. This has 11 subscales and higher scores are indicative of good outcomes.
5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC) (Arms C & D) | Day 1 & Day 8
  The 5D-ASC consists of a set of 94 items that participants are asked to rate to what extent the statements apply to one's particular experience, compared to normal waking consciousness. This has 11 subscales and higher scores are indicative of good outcomes.
5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC) (Arm E) | Day 1, Day 8, & Day 15
  The 5D-ASC consists of a set of 94 items that participants are asked to rate to what extent the statements apply to one's particular experience, compared to normal waking consciousness. This has 11 subscales and higher scores are indicative of good outcomes.
Hallucinogen Rating Scale (HRS) (Arms A & B) | Day 1 & Day 22
  The HRS is a questionnaire with up to 100 items and is designed to assess the subjective effects of hallucinogenic substances. Responses to the majority of questions are on a 5 point intensity scale: 0=not at all; 1=slightly; 2=moderately; 3=quite a bit; and 4=extremely. Some questions have a slightly modified scale, and one question asks to rate the amount of time between when the drug was administered and feeling an effect from: no effect, 0 5 minutes, 5-15 minutes, 15-30 minutes, 30 60 minutes, or more than one hour. The minimum score is zero and maximum score is 400 with higher scores indicating greater hallucinogenic effect.
Hallucinogen Rating Scale (HRS) (Arms C & D) | Day 1 & Day 8
  The HRS is a questionnaire with up to 100 items and is designed to assess the subjective effects of hallucinogenic substances. Responses to the majority of questions are on a 5 point intensity scale: 0=not at all; 1=slightly; 2=moderately; 3=quite a bit; and 4=extremely. Some questions have a slightly modified scale, and one question asks to rate the amount of time between when the drug was administered and feeling an effect from: no effect, 0 5 minutes, 5-15 minutes, 15-30 minutes, 30 60 minutes, or more than one hour. The minimum score is zero and maximum score is 400 with higher scores indicating greater hallucinogenic effect.
Hallucinogen Rating Scale (HRS) (Arm E) | Day 1, Day 8, & Day 15
  The HRS is a questionnaire with up to 100 items and is designed to assess the subjective effects of hallucinogenic substances. Responses to the majority of questions are on a 5 point intensity scale: 0=not at all; 1=slightly; 2=moderately; 3=quite a bit; and 4=extremely. Some questions have a slightly modified scale, and one question asks to rate the amount of time between when the drug was administered and feeling an effect from: no effect, 0 5 minutes, 5-15 minutes, 15-30 minutes, 30 60 minutes, or more than one hour. The minimum score is zero and maximum score is 400 with higher scores indicating greater hallucinogenic effect.
Persisting Effects Questionnaire (PEQ) (Arms A & B) | Day 1 & Day 22
  The PEQ is a 5-item questionnaire that assesses the meaningfulness, spiritual significance, psychological insightfulness, and how psychologically challenging a participant experience was during the medicine session. Scores are assessed on a scale from 0 (not at all) to 5 (extremely). Higher scores (under consideration of reverse-scored items) indicate stronger persisting treatment effects.
Persisting Effects Questionnaire (PEQ) (Arms C & D) | Day 1 & Day 8
  The PEQ is a 5-item questionnaire that assesses the meaningfulness, spiritual significance, psychological insightfulness, and how psychologically challenging a participant experience was during the medicine session. Scores are assessed on a scale from 0 (not at all) to 5 (extremely). Higher scores (under consideration of reverse-scored items) indicate stronger persisting treatment effects.
Persisting Effects Questionnaire (PEQ) (Arm E) | Day 1, Day 8, & Day 15
  The PEQ is a 5-item questionnaire that assesses the meaningfulness, spiritual significance, psychological insightfulness, and how psychologically challenging a participant experience was during the medicine session. Scores are assessed on a scale from 0 (not at all) to 5 (extremely). Higher scores (under consideration of reverse-scored items) indicate stronger persisting treatment effects.
VAS Ratings of "Any Drug Effect" (Arms A & B) | Day 1 & Day 22
  The visual analog scale (VAS) for "Any Drug Effect" consists of a 100mm bipolar line with the far-left side of the line marked "not at all" and the far-right side of the line marked "extremely" to assess if participants feel any drug effect.
VAS Ratings of "Any Drug Effect" (Arms C & D) | Day 1 & Day 8
  The visual analog scale (VAS) for "Any Drug Effect" consists of a 100mm bipolar line with the far-left side of the line marked "not at all" and the far-right side of the line marked "extremely" to assess if participants feel any drug effect.
VAS Ratings of "Any Drug Effect" (Arm E) | Day 1, Day 8, & Day 15
  The visual analog scale (VAS) for "Any Drug Effect" consists of a 100mm bipolar line with the far-left side of the line marked "not at all" and the far-right side of the line marked "extremely" to assess if participants feel any drug effect.
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score from screening (Arms A & B) | Screening, Day -1, Day 1, Day 10, Day 17, Day 31, & Day 38
  The minimum and maximum values are 0 and 60 with a higher score indicating a worse outcome.
Pharmacokinetic parameter of psilocin (Cmax) (Arms A & B) | Day 1, Day 2, Day 22, & Day 23
  Cmax: maximum concentration of plasma psilocin determined from concentrations-versus-time data.
Pharmacokinetic parameter of psilocin (Cmax) (Arms C & D) | Day 1, Day 2, Day 8, & Day 9
  Cmax: maximum concentration of plasma psilocin determined from concentrations-versus-time data.
Pharmacokinetic parameter of psilocin (Cmax) (Arm E) | Day 1, Day 2, Day 8, Day 9, Day 15, & Day 16
  Cmax: maximum concentration of plasma psilocin determined from concentrations-versus-time data.
Pharmacokinetic parameter of psilocin (AUC) (Arms A & B) | Day 1, Day 2, Day 22, & Day 23
  AUC: Area under the plasma concentrations-versus-time curve determined using the linear trapezoidal rule.
Pharmacokinetic parameter of psilocin (AUC) (Arms C & D) | Day 1, Day 2, Day 8, & Day 9
  AUC: Area under the plasma concentrations-versus-time curve determined using the linear trapezoidal rule.
Pharmacokinetic parameter of psilocin (AUC) (Arm E) | Day 1, Day 2, Day 8, Day 9, Day 15, & Day 16
  AUC: Area under the plasma concentrations-versus-time curve determined using the linear trapezoidal rule.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Inamdar, MBBS,DNB,MFPM, Study Director — Cybin IRL Limited
Locations (3):
- United States (3):
  - CenExel ACMR, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: New Jersey Site Recruitment Website. Please click on link to apply — http://depressionpsychedelicstudy.com